CLINICAL TRIAL: NCT07254065
Title: Starting Early to Prevent Obesity Using Telehealth (StEP OUT): Pilot RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-1078 Aim 3; K23HL159326 (NIH)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Feasibility and Acceptability; Prevention Childhood Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- StEP OUT (Experimental): Online nutrition education and parenting support with group chat.
  Interventions: Behavioral: StEP OUT
- Infant Safety Education (Active Comparator): Periodic text messages with links to prenatal and infant health and safety resources.
  Interventions: Behavioral: Infant Safety Education

INTERVENTIONS:
Behavioral: StEP OUT — The program consists of five interactive, virtual, group sessions (two prenatal, three post-natal) with a registered dietician/lactation counselor and other women/families of similar gestational age/infant age. Participants discuss maternal nutrition, responsive feeding techniques (breast and bottle), infant feeding cues, and non-feeding soothing methods. Participants are also invited to participate in a moderated WhatsApp Chat with each other to foster additional social engagement and connection. They participate in the program until the baby turns 6 months.
  Arms: StEP OUT
Behavioral: Infant Safety Education — This intervention consists of periodic text messages (approximately every 2 weeks) with links to prenatal health and infant safety information.
  Arms: Infant Safety Education

SUMMARY:
The goal of this clinical trial is to test an online program that teaches healthy habits during pregnancy and infant to prevent early child obesity in Latino families. Specifically, this pilot trial will determine how well we can deliver and test the effects of the program, and how acceptable it is to participants.

The main question it aims to answer are:

• Is a randomized controlled trial of StEP OUT versus infant safety education control feasible to conduct and acceptable to participants? Researchers will compare StEP OUT to infant safety education control to see if participants enroll in and engage with the program, complete surveys, and learn the content we are teaching.

Participants will:

* Be assigned to receive StEP OUT or Infant Safety Education
* If receiving StEP OUT, they will participant in group text chats and video calls
* If receiving Infant Safety Education, they will receive periodic text messages with helpful links and tips
* Respond to periodic surveys

DETAILED DESCRIPTION:
Our objective is to conduct a pilot RCT to evaluate the acceptability, feasibility, and preliminary effectiveness of StEP OUT.

Hypothesis: The intervention and control conditions of StEP OUT will be acceptable to families and feasible, as measured by recruitment, randomization, retention, usability, and fidelity. H3b (exploratory): Families exposed to StEP OUT will have improved obesity-related outcomes (knowledge, styles, practices, and infant adiposity) compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with singleton of 24 to 32 weeks estimated gestational age
* Self-identify as Hispanic/Latinx
* Speak fluent English or Spanish
* At least 18 years of age
* Has a phone or device to participate in video calls
* Receiving or eligible to receive New York State Medicaid benefits

Exclusion Criteria:

* Diminished mental capacity
* Serious medical or psychiatric illness
* Fetal condition expected to substantially influence infant feeding (anatomic abnormality, such as cleft lip/palate or one that will require surgery within the first six months of life, chromosomal abnormality, such as Down's syndrome or other trisomy, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability | From enrollment through the end of the study after child age 6 months
  We will use the Sekhon acceptability framework to assess affective attitude, burden, opportunity cost, perceived effectiveness, coherence, ethicality, self-efficacy and general acceptability.

SECONDARY OUTCOMES:
Feasibility | From enrollment to study completion after infant age 6 months.
  Feasibility assessment will include measures of recruitment (number enrolled of those eligible), retention (number who attend all scheduled sessions of those enrolled), fidelity (number of curriculum components delivered of those planned), and attendance (1. Attendance rate: number of participants who attend each sessions of those scheduled to attend; 2. Program dose: number of sessions attended for each participant)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD underlying the primary outcomes will be shared. Sensitive variables (e.g., location-based identifiers, audio/video files, free-text fields) will not be shared. A data dictionary, protocol, and SAP will be provided.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available beginning 12 months after publication for 5 years.
Access Criteria: Access requires a proposal and a data use agreement.